CLINICAL TRIAL: NCT06778174
Title: Prospective Analysis of the Treatment of Progressive Familial Intrahepatic Cholestasis (TreatFIC)
Acronym: TreatFIC
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Henkjan J. Verkade, Pediatric hepatologist, Professor of pediatrics, University Medical Center Groningen
Other Study IDs: UGroningen - PaNaMaID11162
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Progressive Familial Intrahepatic Cholestasis
Keywords: PFIC; ASBT; IBAT; biliary diversion; liver transplantation
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1 | interventions — Observation; Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- FIC1-deficiency: genetically proven deficiency of FIC1 (FIC1). Disease is also known as PFIC1.
  Interventions: Other: observational study
- BSEP-deficiency: genetically proven deficiency of Bile Salt Export Pump (BSEP, ABCB11). Disease is also known as PFIC2.
  Interventions: Other: observational study
- MDR3-deficiency: genetically proven deficiency of Multi Drug Resistance protein type 3 (MDR3, ABCB4). Disease is also known as PFIC3.
  Interventions: Other: observational study
- Other genetic subtypes of Familiai Intrahepatic Cholestasis: TJP2 deficiency (TJP2), FXR deficiency (NR1H4), SLC51A deficiency (SLC51A), USP53 deficiency (USP53), KIF12 deficiency (KIF12), ZFYE19 deficiency (ZFYVE19), MYO5B deficiency (MYO5B), SEMA7A deficiency (SEMA7A), VPS33B deficiency, (VPS33B), PSKH1 deficiency (PSKH1)
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — The interventions are not determined by the study, which is purely observational on "real world data".
  Other Names: natural history; surgical biliary diversion; liver transplantation; IBAT-inhibition

SUMMARY:
The project has the following general aims:

1. Natural course and prognosis: To prospectively follow the natural course and prognosis of the different types of PFIC, to broaden the understanding of the different very rare diseases and to allow predictions about the course of disease in different types of PFIC.
2. Efficacy: To define the course of disease in FIC patients and identify associations with different treatments (symptomatic treatments, interruption of the enterohepatic circulation by surgical or medical means and other therapies such as corrector/potentiator or exon skipping therapy. The course of disease will be characterized by biochemical, clinical and surgical parameters, including liver transplantation.
3. Safety: To define the complications associated with the different treatments (symptomatic treatments, interruption of the enterohepatic circulation by surgical or medical means and other therapies such as corrector/potentiator or exon skipping therapy, liver transplantation). Follow up will be as long as possible.
4. (Surrogate) biomarker response: Biochemical parameters will be longitudinally collected and associated with changes in treatments / course of disease.
5. Genotype-phenotype relationships: If patient numbers permit, to establish genotype-phenotype relationships for (non)responsiveness towards different treatments in patients with genetic mutations causing the different forms of FIC disease.

ELIGIBILITY:
Inclusion Criteria:

- Genetically confirmed cases of a PFIC type disease: FIC1 deficiency, BSEP deficiency, MDR3 deficiency, TJP2 deficiency, FXR deficiency, SLC51A deficiency, USP53 deficiency, KIF12 deficiency, ZFYE19 deficiency, MYO5B deficiency, SEMA7A deficiency, VPS33B deficiency, PSKH1 deficiency.

Exclusion Criteria:

- Cases with suspected PFIC type disease, but without genetic testing data available.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The diagnosis of a PFIC type disease needs to be performed according to the international guidelines, based on (episodes with a) low gamma-GT cholestasis and identification of disease-causing mutations in the indicated genes.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with liver transplantation | at 5, 10, 15 and 18 years of age, as well as >18 years of age
  The number (percentage) of patients undergoing liver transplantation related to the age of the patient

SECONDARY OUTCOMES:
Number of participants that succumbed | at 5, 10, 15 and 18 years of age, as well as >18 years of age
  Mortality related to age of the patient

OTHER OUTCOMES:
Number of participant undergoing a surgical biliary diversion | at 5, 10, 15 and 18 years of age, as well as >18 years of age
  Number of participant undergoing a surgical biliary diversion related to age

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Ownership of individal patient data will remain in the hands of the participating centers.

REFERENCES:
- [Background] Felzen A, Verkade HJ. The spectrum of Progressive Familial Intrahepatic Cholestasis diseases: Update on pathophysiology and emerging treatments. Eur J Med Genet. 2021 Nov;64(11):104317. doi: 10.1016/j.ejmg.2021.104317. Epub 2021 Aug 31. PMID 34478903
- [Background] Felzen A, van Wessel DBE, Gonzales E, Thompson RJ, Jankowska I, Shneider BL, Sokal E, Grammatikopoulos T, Kadaristiana A, Jacquemin E, Spraul A, Lipinski P, Czubkowski P, Rock N, Shagrani M, Broering D, Nicastro E, Kelly D, Nebbia G, Arnell H, Fischler B, Hulscher JBF, Serranti D, Arikan C, Polat E, Debray D, Lacaille F, Goncalves C, Hierro L, Munoz Bartolo G, Mozer-Glassberg Y, Azaz A, Brecelj J, Dezsofi A, Calvo PL, Grabhorn E, Hartleif S, van der Woerd WJ, Kamath BM, Wang JS, Li L, Durmaz O, Kerkar N, Jorgensen MH, Fischer R, Jimenez-Rivera C, Alam S, Cananzi M, Laverdure N, Ferreira CT, Guerrero FO, Wang H, Sency V, Kim KM, Chen HL, de Carvalho E, Fabre A, Bernabeu JQ, Zellos A, Alonso EM, Sokol RJ, Suchy FJ, Loomes KM, McKiernan PJ, Rosenthal P, Turmelle Y, Horslen S, Schwarz K, Bezerra JA, Wang K, Hansen BE, Verkade HJ; NAtural course and Prognosis of PFIC and Effect of biliary Diversion (NAPPED) Consortium. Genotype-phenotype relationships of truncating mutations, p.E297G and p.D482G in bile salt export pump deficiency. JHEP Rep. 2022 Nov 16;5(2):100626. doi: 10.1016/j.jhepr.2022.100626. eCollection 2023 Feb. PMID 36687469
- [Background] van Wessel DBE, Gonzales E, Hansen BE, Verkade HJ. Defining the natural history of rare genetic liver diseases: Lessons learned from the NAPPED initiative. Eur J Med Genet. 2021 Jul;64(7):104245. doi: 10.1016/j.ejmg.2021.104245. Epub 2021 May 13. PMID 33991701
- [Background] van Wessel DBE, Thompson RJ, Gonzales E, Jankowska I, Shneider BL, Sokal E, Grammatikopoulos T, Kadaristiana A, Jacquemin E, Spraul A, Lipinski P, Czubkowski P, Rock N, Shagrani M, Broering D, Algoufi T, Mazhar N, Nicastro E, Kelly D, Nebbia G, Arnell H, Fischler B, Hulscher JBF, Serranti D, Arikan C, Debray D, Lacaille F, Goncalves C, Hierro L, Munoz Bartolo G, Mozer-Glassberg Y, Azaz A, Brecelj J, Dezsofi A, Luigi Calvo P, Krebs-Schmitt D, Hartleif S, van der Woerd WL, Wang JS, Li LT, Durmaz O, Kerkar N, Horby Jorgensen M, Fischer R, Jimenez-Rivera C, Alam S, Cananzi M, Laverdure N, Targa Ferreira C, Ordonez F, Wang H, Sency V, Mo Kim K, Chen HL, Carvalho E, Fabre A, Quintero Bernabeu J, Alonso EM, Sokol RJ, Suchy FJ, Loomes KM, McKiernan PJ, Rosenthal P, Turmelle Y, Rao GS, Horslen S, Kamath BM, Rogalidou M, Karnsakul WW, Hansen B, Verkade HJ; Natural Course and Prognosis of PFIC and Effect of Biliary Diversion Consortium. Impact of Genotype, Serum Bile Acids, and Surgical Biliary Diversion on Native Liver Survival in FIC1 Deficiency. Hepatology. 2021 Aug;74(2):892-906. doi: 10.1002/hep.31787. Epub 2021 Jul 13. PMID 33666275
- [Background] van Wessel DBE, Thompson RJ, Gonzales E, Jankowska I, Sokal E, Grammatikopoulos T, Kadaristiana A, Jacquemin E, Spraul A, Lipinski P, Czubkowski P, Rock N, Shagrani M, Broering D, Algoufi T, Mazhar N, Nicastro E, Kelly DA, Nebbia G, Arnell H, Bjorn Fischler, Hulscher JBF, Serranti D, Arikan C, Polat E, Debray D, Lacaille F, Goncalves C, Hierro L, Munoz Bartolo G, Mozer-Glassberg Y, Azaz A, Brecelj J, Dezsofi A, Calvo PL, Grabhorn E, Sturm E, van der Woerd WJ, Kamath BM, Wang JS, Li L, Durmaz O, Onal Z, Bunt TMG, Hansen BE, Verkade HJ; NAtural course and Prognosis of PFIC and Effect of biliary Diversion (NAPPED) consortium. Genotype correlates with the natural history of severe bile salt export pump deficiency. J Hepatol. 2020 Jul;73(1):84-93. doi: 10.1016/j.jhep.2020.02.007. Epub 2020 Feb 20. PMID 32087350